CLINICAL TRIAL: NCT01139970
Title: A Phase I Study of the PARP Inhibitor ABT-888 in Combination With Temozolomide in Acute Leukemias
Brief Title: Veliparib and Temozolomide in Treating Patients With Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01457; NCI-2011-01457 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000674355; GCC 0940; JHUJ1051; JHUJ1051; GCC 0940 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8456 (Other: CTEP); N01CM00071 (NIH); N01CM62201 (NIH); N01CM62209 (NIH); P30CA006973 (NIH); U01CA062487 (NIH); U01CA062502 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p21.3;q23.3); MLLT3-KMT2A; Adult Acute Promyelocytic Leukemia With t(15;17)(q24.1;q21.2); PML-RARA; Adult B Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Adult T Acute Lymphoblastic Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Chronic | interventions — Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (temozolomide and veliparib) (Experimental): Patients receive veliparib PO QD on day 1 and twice daily on days 4-12 and temozolomide PO QD on days 3-9 of course 1.
  Beginning at least 30 days after the start of treatment, patients receive veliparib PO BID on days 1-8 and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients achieving complete remission receive 5 more courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temozolomide; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I clinical trial is studies the side effects and best dose of giving veliparib together with temozolomide in treating patients with acute leukemia. Veliparib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving veliparib together with temozolomide may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum-tolerated dose (MTD) and recommended phase II dose of ABT-888 (veliparib) administered in combination with temozolomide in patients with acute leukemias.

II. To evaluate the feasibility, safety, and toxicity of administering ABT-888 in combination with temozolomide in patients with acute leukemias.

SECONDARY OBJECTIVES:

I. To document response in acute leukemias. II. To observe the pharmacokinetics of both ABT-888 and temozolomide when administered alone and in combination.

III. To study the pharmacodynamics to determine the levels of poly(ADP-ribose) (PAR) before and after administration of ABT-888 and temozolomide in patient leukemia blasts, to analyze methyl-guanine methyl-transferase (MGMT) protein levels in primary leukemia blasts, and to quantify the induction of gamma-H2A histone family, member X (y-H2AX) and RAD51 recombinase (RAD51) foci in patient leukemia blasts after treatment.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib orally (PO) once daily (QD) on day 1 and twice daily on days 4-12 and temozolomide PO QD on days 3-9 of course 1.

Beginning at least 30 days after the start of treatment, patients receive veliparib PO twice daily (BID) on days 1-8 and temozolomide PO QD on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients achieving complete remission receive 5 more courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of one of the following:

  * Relapsed or refractory acute myeloid leukemia (AML); patients with acute promyelocytic leukemia t(15;17) must have failed tretinoin (ATRA), arsenic, and gemtuzumab ozogamycin to be eligible (patients should be refractory to all three agents-absence of durable hematologic response or relapse with complete remission [CR] duration of less than 6 months)
  * Relapsed or refractory pre-B- or T-cell acute lymphoblastic leukemia (ALL); patients with Philadelphia chromosome-positive (Ph+) ALL [t(9;22)] will be eligible provided that they have failed (intolerance/resistance) at least 2 different tyrosine kinase inhibitors (TKIs) or have a mutation associated with resistance to TKIs (T315I)
  * Chronic myelogenous leukemia (CML) in accelerated or blastic phase; patients failed (resistance/intolerance) at least 2 different TKIs or have a mutation associated with resistance to TKIs (T315I)
  * Chronic myelomonocytic leukemia-2 (CMML-2) defined as having > 10% blasts (including promonocytes) in the bone marrow or > 5-19% blasts (including promonocytes) in the peripheral blood
  * AML arising in the setting of antecedent myelodysplasia (MDS) or myeloproliferative disorder (MPD)
  * Therapy-related AML
  * Untreated AML in adults 60 years of age and older who are not candidates for induction chemotherapy due to poor-risk features including adverse cytogenetics or molecular markers (fms-related tyrosine kinase 3 [FLT3] internal tandem duplication [ ITD]+), or are unwilling to receive intensive induction chemotherapy; adverse cytogenetics: complex karyotype (>= 3 chromosomal abnormalities), 5q-, 7q-, 9q-, 20q-, abn12p, +21, +8, t(6;9), t(6;11), t(11;19), -7, -5, inv3/t(3;3), abn11q23, abn17p, abn21q
  * Untreated ALL in adults 60 years of age and older who are not candidates for induction chemotherapy due to poor-risk features including adverse cytogenetics [t(4;11); t(1;19), hypodyploidy] or are unwilling to receive intensive induction chemotherapy; patients with Ph+ ALL [t(9;22)] will be eligible provided that they have failed (intolerance/resistance) at least 2 different TKIs or have a mutation associated with resistance to TKIs (T315I)
* Previous therapy

  * Only patients who have received or are ineligible for established curative regimens, including stem cell transplantation when applicable, can be enrolled on this study
  * Patients may have received any number of prior chemotherapy regimens, which may include allogeneic or autologous transplantation, provided that performance status and organ function are maintained
  * Previous cytotoxic chemotherapy should have been completed at least 3 weeks and radiotherapy at least 2 weeks prior to treatment on the study (6 weeks if the last regimen included carmustine [BCNU] or mitomycin C) and all adverse events (excluding alopecia, acne, rash) due to agents administered more than 3 weeks earlier should recover to =< grade 1; patients with hematologic malignancies are expected to have hematologic abnormalities at study entry; these abnormalities which are thought to be primarily related to the underlying leukemia, are not considered to be toxicities (AE) and do not need to resolve to =< grade 1
  * Patients should stop taking all biologic agents including hematopoietic growth factors, imatinib or similar TKIs, at least 1 week prior to treatment on the study and all adverse events (excluding alopecia, acne, rash) due to agents administered more than 1 week earlier should recover to =< grade 1; since only patients with advanced Ph+ ALL and CML in accelerated/blast phase are eligible for this study, this short period off TKIs was selected to avoid rapid leukemia progression; if using hydroxyurea, corticosteroids, or leukopheresis for blast count control, patients must be off >= 24 hrs before starting treatment on the study
  * Patients who have undergone autologous stem cell transplantation (ASCT) are eligible provided that they are >= 4 weeks from stem cell infusion and meet other eligibility criteria
  * Patients who have undergone allogeneic SCT (alloSCT) are eligible if they are >= 60 days post stem cell infusion, have no evidence of graft vs. host disease, and are >= 2 weeks off all immunosuppressive therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients have to be able to swallow pills
* Total or direct bilirubin < 2 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 5 X institutional upper limit of normal
* Creatinine < 2 mg/dl
* Female patients of childbearing potential must have a negative pregnancy test
* Female patients of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days afterward; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents, or concurrent chemotherapy, radiation therapy, or immunotherapy
* Any previous treatment with temozolomide
* Patients with active central nervous system leukemia are excluded from this clinical trial because they may develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; patients with a history of central nervous system (CNS) leukemia but no active disease at the time of enrollment are eligible
* Hyperleukocytosis with > 30,000 blasts/ul; (if using hydroxyurea, corticosteroids, or leukopheresis for blast count control, patients must be off >= 24 hrs before starting treatment on the study); once patient starts treatment on the study the hydroxyurea use should be avoided, however, for patients with rapidly proliferating disease use of hydroxyurea is allowed on treatment days 1 through 12 if it becomes necessary to control a rising white blood cell (WBC) or leukostasis; the WBC need not reach 30,000/ul to start hydroxyurea during protocol days 1-12; the decision to start hydroxyurea during this time is at the discretion of the treating physician
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or temozolomide used in this study
* Active, uncontrolled infection; patients with infection under active treatment and controlled with antibiotics are eligible
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ABT-888
* Known human immunodeficiency virus (HIV) infected patients (HIV testing will not be performed as a part of screening) on combination antiretroviral therapy, exclusive of zidovudine or starvudine, or HIV infected patients not on or willing to suspend antiretroviral therapy will be eligible provided that their cluster of differentiation (CD)4 cell count is greater than 250/mm3; HIV infected patients with CD4 count equal or less than 250/mm3 will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-06-04 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
MTD of veliparib, determined according to incidence of dose limiting toxicity, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 28 days

SECONDARY OUTCOMES:
Response rate at the MTD, assessed using revised International Working Group response criteria | Up to 30 days
  The proportion of responders will be estimated and reported with the corresponding 90% confidence interval.
Changes in levels of poly(ADP-ribose) (PAR) | From baseline to 6 hours after drug administration on day 1 of course 1
  The proportion of subjects with significant inhibition will be estimated for each dose level. Summary statistics and results of the statistical tests for contingency tables will be reported.
Average expression of MGMT | Up to 30 days
  Average expression of MGMT will be measured and classified as positive versus negative (less than 20% of mean value) for all patients regardless of the administered drug dose. We will use the Fisher's exact test for 2 x 2 tables to assess whether the lack of MGMT expression correlates with the response.
Average change from baseline level in y-H2AX foci | From baseline to 30 days
  The average change from baseline level in γ-H2AX and RAD51 foci will be estimated for all patients to assess whether increase in foci and response to treatment are associated. Assessed using a single group repeated measures analysis of variance (ANOVA) with 0.05 significance level.
Average change from baseline level in RAD51 foci | From baseline to 30 days
  The average change from baseline level in γ-H2AX and RAD51 foci will be estimated for all patients to assess whether increase in foci and response to treatment are associated. Assessed using a single group repeated measures ANOVA with 0.05 significance level.
Non-homologous end joining repair | Up to 30 days
  Repeated measures data structure will provide adequate power to estimate intra- and inter-patient variability.
Double strand break (DSB) repair | Up to 30 days
  The plausible relationship between change in DSB repair and clinical response will be examined using the Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (3):
- United States (3):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland